CLINICAL TRIAL: NCT01021813
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Long Term Safety Study of MK-4305 in Patients With Primary Insomnia
Brief Title: A Long Term Safety Study of Suvorexant in Participants With Primary Insomnia (MK-4305-009 AM3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-009; 2009_696 (Other: Merck Registration Number)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suvorexant (Experimental): After a 1-week single-blind placebo run-in, participants received suvorexant (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime for 12 months during the Treatment Phase.
  Interventions: Drug: Suvorexant; Drug: Dose-matched Placebo to Suvorexant
- Placebo (Placebo Comparator): After a 1-week single-blind placebo run-in, participants received dose-matched placebo to suvorexant (administered according to age) daily before bedtime for 12 months during the Treatment Phase.
  Interventions: Drug: Dose-matched Placebo to Suvorexant

INTERVENTIONS:
Drug: Suvorexant — Oral tablet (30 mg and 10 mg), administered daily before bedtime
  Other Names: MK-4305
  Arms: Suvorexant
Drug: Dose-matched Placebo to Suvorexant — Oral tablet, administered daily before bedtime

SUMMARY:
This study will establish the safety and tolerability of suvorexant (MK-4305) when administered for up to 14 months. Participants will be randomized to receive suvorexant or placebo for a 12-month double-blind (DB) Treatment Phase. Participants who complete the 12-month DB Treatment Phase will enter a 2-month DB Randomized Discontinuation Phase. At the time of initial randomization, participants assigned to receive suvorexant during the initial 12-month Treatment Phase will be simultaneously randomized, in a 1:1 ratio, to receive either suvorexant or placebo during the 2-month Randomized Discontinuation Phase. Participants randomized to receive placebo in the initial 12-month Treatment Phase will continue to receive placebo during the 2-month Randomized Discontinuation Phase.

The first 3 nights of the Randomized Discontinuation Phase are referred to as the Run-Out Phase, and will assess rebound and withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia
* Participant is able to read, understand, and complete questionnaires and diaries
* If female, participant and partner both agree to use acceptable contraception. If male partner does not use an effective form of contraception, female participant must use 2 acceptable forms of contraception
* If ≥65 years of age, score of ≥25 on the Mini Mental State Examination (MMSE)

Exclusion Criteria:

* If female, participant is pregnant
* Participant expects to donate eggs or sperm during the study
* Recent and/or active history of a confounding neurological disorder
* History of clinically unstable cardiovascular disorder within the last 6 months
* Lifetime history of bipolar disorder
* Psychiatric condition that requires treatment with a medication prohibited by the study, or any other psychiatric condition that would interfere with the participant's ability to participate in the study
* History of substance abuse/dependence
* History of cancer ≤5 years prior to study participation except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Evidence of suicidality (based on a score of 2 on the Quick Inventory of Depressive Symptomatology Self-Report 16-Item ([QIDS-SR16] suicide item #12)
* Participant has travelled across >3 time zones or >3 hour time difference in the last 2 weeks
* History of permanent night shift work or rotating day/night shift work in the past 2 weeks
* Body Mass Index (BMI) >40 kg/m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2009-12-10 (Actual); Primary Completion 2011-05-17 (Actual); Study Completion 2011-08-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Suvorexant in Elderly Patients with Insomnia: Pooled Analyses of Data from Phase III Randomized Controlled Clinical Trials. Am J Geriatr Psychiatry. 2017 Jul;25(7):791-802. doi: 10.1016/j.jagp.2017.03.004. Epub 2017 Mar 8. PMID 28427826
- [Derived] Herring WJ, Connor KM, Snyder E, Snavely DB, Zhang Y, Hutzelmann J, Matzura-Wolfe D, Benca RM, Krystal AD, Walsh JK, Lines C, Roth T, Michelson D. Clinical profile of suvorexant for the treatment of insomnia over 3 months in women and men: subgroup analysis of pooled phase-3 data. Psychopharmacology (Berl). 2017 Jun;234(11):1703-1711. doi: 10.1007/s00213-017-4573-1. Epub 2017 Mar 7. PMID 28265715
- [Derived] Michelson D, Snyder E, Paradis E, Chengan-Liu M, Snavely DB, Hutzelmann J, Walsh JK, Krystal AD, Benca RM, Cohn M, Lines C, Roth T, Herring WJ. Safety and efficacy of suvorexant during 1-year treatment of insomnia with subsequent abrupt treatment discontinuation: a phase 3 randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 May;13(5):461-71. doi: 10.1016/S1474-4422(14)70053-5. Epub 2014 Mar 27. PMID 24680372
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-009&kw=4305-009&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 781 participants randomized into the Treatment Phase, 522 were randomized to suvorexant and 259 were randomized to placebo. Two participants were randomized, but not treated (one from each treatment group); therefore, the total number of participants evaluated for safety was 779.
Groups:
- Suvorexant: After a 1-week single-blind placebo run-in, participants received suvorexant (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime for 12 months during the double-blind (DB) Treatment Phase.
- Placebo: After a 1-week single-blind placebo run-in, participants received dose-matched placebo to suvorexant (administered according to age) daily before bedtime for 12 months during the DB Treatment Phase.
- Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation): Following treatment with suvorexant during the 12-Month DB Treatment Phase, participants received their same dose of suvorexant during a 2-month DB Randomized Discontinuation Phase.
- Suvorexant (DB Treatment)/Placebo (DB Discontinuation): Following treatment with suvorexant during the 12-Month DB Treatment Phase, participants received dose-matched placebo to suvorexant during a 2-month DB Randomized Discontinuation Phase.
- Placebo (DB Treatment)/Placebo (DB Discontinuation): Following treatment with dose-matched placebo to suvorexant during the 12-Month DB Treatment Phase, participants continued to receive dose-matched placebo to suvorexant during a 2-month DB Randomized Discontinuation Phase.
Period: DB Treatment Phase
Arm/Group | Suvorexant | Placebo | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation)
Started | 522 | 259 | 0 | 0 | 0
Treated | 521 | 258 | 0 | 0 | 0
Completed | 322 | 162 | 0 | 0 | 0
Not Completed | 200 | 97 | 0 | 0 | 0
Not completed — Adverse Event | 60 | 22 | 0 | 0 | 0
Not completed — Lack of Efficacy | 44 | 28 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 12 | 0 | 0 | 0
Not completed — Physician Decision | 17 | 8 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 60 | 24 | 0 | 0 | 0
Period: DB Randomized Discontinuation Phase
Arm/Group | Suvorexant | Placebo | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation)
Started | 0 | 0 | 156 | 166 | 162
Completed | 0 | 0 | 152 | 161 | 157
Not Completed | 0 | 0 | 4 | 5 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: 781 participants were randomized on study (suvorexant=522, placebo=259). 2 participants were randomized but not treated, thus the total number of participants evaluated for baseline age and gender was 779 (suvorexant=521, placebo=258). 771 participants had data available for evaluation of baseline sleep parameters (suvorexant=517, placebo=254)
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 521 | 258 | 779
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.5) | 62.0 (14.6) | 61.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 149 | 436
  Male | 234 | 109 | 343
Mean Subjective Total Sleep Time (sTSTm) [Mean (Standard Deviation); unit: minutes] — The baseline sTSTm was defined as the participant's reported total amount of time spent asleep before waking for the day (measured in minutes), calculated as the mean of the last 7 (non-missing) daily e-diary values obtained during the placebo run-in phase.
  (n=517, n=254)
  minutes | 320.4 (76.1) | 329.9 (79.4) | 323.5 (77.3)
Mean Subjective Time to Sleep Onset in minutes (sTSOm) [Mean (Standard Deviation); unit: minutes] — The baseline sTSOm was defined as the participant's reported time that he or she required to fall asleep (measured in minutes), calculated as the mean of the last 7 (non-missing) daily e-diary values obtained during the placebo run-in phase.
  (n=517, n=254)
  minutes | 65.9 (63.8) | 65.0 (60.6) | 65.6 (62.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Cataplexy Adverse Events (AEs) During the Double-Blind (DB) Treatment Phase
Description: Cataplexy is defined as a sudden loss of muscle tone while awake which prevents voluntary movement.
Time Frame: From the first day of study treatment up to 12 months
Population: All Participants as Treated (APaT) population; all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants Who Experienced Sleep Paralysis AEs During the DB Treatment Phase
Description: Sleep paralysis was defined as the inability to perform voluntary muscle movements during sleep. Sleep paralysis adverse events included sleep-onset paralysis (paralysis as one is falling asleep).
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants | 0.4 | 0.0
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to construct the confidence interval for the difference in the percentage of participants with any sleep paralysis AEs between the Suvorexant group and Placebo group; Test type: Superiority or Other; Miettinen & Nurminen Method; Difference in Percentage = 0.4, 95% CI 2-sided [-1.1 to 1.4]

3. Primary Outcome: Percentage of Participants Who Experienced Complex Sleep-related Behaviors AEs During the DB Treatment Phase
Description: Complex sleep-related behaviors were reported as ECIs and were characterized by patients engaging in specific activities while asleep (e.g., eating, drinking, preparing meals, making phone calls, having sex, driving, and sleep walking).
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants
  any complex sleep-related behaviors | 0.2 | 0.0
  somnambulism | 0.2 | 0.0
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to construct the confidence interval for the difference in the percentage of participants with any complex sleep-related behaviors AEs between the Suvorexant group and Placebo group; Test type: Superiority or Other; p = 0.482, Miettinen & Nurminen Method; Difference in Percentage = 0.2, 95% CI 2-sided [-1.3 to 1.1]

4. Primary Outcome: Percentage of Participants Who Experienced Falls AEs During the DB Treatment Phase
Description: Falls were adjudicated (to establish whether a fall event was due to cataplexy).
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants | 2.3 | 3.1
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to calculate the p-value and construct the confidence interval for the difference in the percentage of participants with any falls AEs between the Suvorexant group and Placebo group; Test type: Superiority or Other; p = 0.508, Miettinen & Nurminen Method; Difference in Percentage = -0.8, 95% CI 2-sided [-3.9 to 1.5]

5. Primary Outcome: Percentage of Participants Who Experienced Suicidal Ideation and/or Behavior AEs During the DB Treatment Phase
Description: Suicidal ideation included suicidal plans, suicidal tendency, death wishes, life weariness, and suicidal intention. Suicidal behaviors included suicide attempts, suicide gesture, and self-injurious behaviour. Suicidal ideation and/or behavior was reported as an AE and considered an ECI.
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants | 0.8 | 0.0
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to calculate the p-value and construct the confidence interval for the difference in the percentage of participants with any suicidal ideation/behavior AEs considered an ECI between the Suvorexant group and Placebo group; Test type: Superiority or Other; p = 0.159, Miettinen & Nurminen Method; Difference in Percentage of AEs = 0.8, 95% CI 2-sided [-0.7 to 2.0]

6. Primary Outcome: Percentage of Participants Who Experienced Hypnagogic/Hypnopompic Hallucinations AEs During the DB Treatment Phase
Description: Perceptual distortions associated with transitions between wakefulness and sleep were termed as hypnagogic (occurring during the onset of sleep) or hypnopompic (occurring during onset of wakefulness) hallucinations.
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants
  Any hypnagogic/hypnopompic hallucinations AEs | 0.8 | 0.0
  Hypnagogic hallucination | 0.6 | 0.0
  Hypnopompic hallucination | 0.2 | 0.0
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to calculate the p-value and construct the confidence interval for the difference in the percentage of participants with any Hypnagogic/hypnopompic hallucinations AEs between the Suvorexant group and Placebo group; Test type: Superiority or Other; p = 0.159, Miettinen & Nurminen Method; Difference in Percentage = 0.8, 95% CI 2-sided [-0.7 to 2.0]

7. Primary Outcome: Percentage of Participants Who Experienced Selected AEs Associated With Potential for Abuse During the DB Treatment Phase
Description: The pre-specified terms which were suggestive of abuse potential on this study included depersonalization (feeling of watching oneself act, while having no control over a situation), derealization (alteration in the perception or experience of the external world so that it seems unreal), dissociation (includes a wide array of experiences from mild detachment from immediate surroundings to more severe detachment from physical and emotional experience), euphoric mood (exaggerated feeling of physical and emotional well-being and optimism not consonant with apparent stimuli or events), mania (state of abnormally elevated or irritable mood, arousal, and/or energy levels), hallucination (perception in the absence of a stimulus which has qualities of real perception), and potential study medication misuse.
Time Frame: From the first day of study treatment up to 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
percentage of participants
  any selected AE of potential abuse | 3.5 | 3.9
  Drug maladministration | 2.3 | 3.9
  Derealisation | 0.2 | 0.0
  Hallucination, auditory | 0.2 | 0.0
  Hallucination, visual | 0.2 | 0.0
  Hypnagogic hallucination | 0.6 | 0.0
  Hypnopompic hallucination | 0.2 | 0.0
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; The method of Miettinen and Nurminen was used to calculate the p-value and construct the confidence interval for the difference in the percentage of participants with any selected AEs associated with potential abuse between the Suvorexant group and Placebo group; Test type: Superiority or Other; p = 0.767, Miettinen & Nurminen Method; Difference in Percentage = -0.4, 95% CI 2-sided [-3.8 to 2.2]

8. Secondary Outcome: Percentage of Participants With Withdrawal Symptoms During the DB Run-Out Phase: Tyrer Withdrawal Symptom Questionnaire (WSQ)
Description: Withdrawal effects assessed using Tyrer WSQ, which evaluated the presence/absence and severity of withdrawal symptoms with 20 items (i.e. sensitivity to noise, light, smell, touch, feeling unreal, etc). The Tyrer WSQ was completed as part of the evening e-diary prior to dosing on the Month 12 visit and on the 3 consecutive evenings of the DB Run-out Phase (first 3 nights of DB Discontinuation Phase). Responses rated 0 (No), 1 (Yes-moderate), or 2 (Yes-severe); range from 0 (no withdrawal) to 40 (severe withdrawal).
  A participant was defined to have a withdrawal symptom if an item during any of the 3 DB Run-out days had emerged for the first time, or had worsened compared to the measurement obtained at the end of the Treatment phase (Month 12). For single night analysis, a patient was defined to have withdrawal effects if the number of withdrawal symptoms (emergent or worsening) was ≥3. For across night analysis, withdrawal was defined as a total of ≥3 symptoms across the 3 nights.
Time Frame: Evening of Month 12 visit and next 3 consecutive days (Night 1, 2, and 3 of Discontinuation Phase [otherwise known as the Run-out])
Population: Participants in the APaT population who completed the entire DB Treatment Phase, had at least one measurement at the end of the DB Treatment Phase (Month 12), had taken at least one dose of Run-out study medication, and had a measurement on at least one of the nights of the DB Run-out Phase.
Measure: Number; unit: percentage of participants
Groups:
- Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation): Following treatment with suvorexant during the 12-Month DB Treatment Period, participants received their same dose of suvorexant during a 2-month DB Discontinuation Period.
- Suvorexant (DB Treatment)/Placebo (DB Discontinuation): Following treatment with suvorexant during the 12-Month DB Treatment Period, participants received dose-matched placebo to suvorexant during a 2-month DB Discontinuation Period.
- Placebo (DB Treatment)/Placebo (DB Discontinuation): Following treatment with dose-matched placebo to suvorexant during the 12-Month DB Treatment Period, participants continued to receive dose-matched placebo to suvorexant during a 2-month DB Discontinuation Period.
Arm/Group | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation)
Number analyzed (Participants) | 129 | 129 | 136
percentage of participants
  Withdrawal Symptoms on Night 1 (n=121, 122, 131) | 0.8 | 1.6 | 1.5
  Withdrawal Symptoms on Night 2 (n=121, 124, 125) | 0.8 | 3.2 | 2.4
  Withdrawal Symptoms on Night 3 (n=116, 120, 128) | 1.7 | 2.5 | 0.8
  Symptoms Across Nights 1, 2, & 3 (n=129, 129, 136) | 6.2 | 6.2 | 5.1
Statistical Analysis 1: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Suvorexant (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with withdrawal symptoms during Night 1 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Suvorexant (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.567, Miettinen & Nurminen Method; Difference in Percentage: Night 1 = -0.81, 95% CI 2-sided [-5.1 to 3.1]
Statistical Analysis 2: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Suvorexant (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with withdrawal symptoms during Night 2 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Suvorexant (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.185, Miettinen & Nurminen Method; Difference in Percentage: Night 2 = -2.40, 95% CI 2-sided [-7.3 to 1.6]
Statistical Analysis 3: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Suvorexant (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with withdrawal symptoms during Night 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Suvorexant (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.680, Miettinen & Nurminen Method; Difference in Percentage: Night 3 = -0.78, 95% CI 2-sided [-5.6 to 3.9]
Statistical Analysis 4: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Suvorexant (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with withdrawal symptoms across Nights 1, 2, and 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Suvorexant (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 1.000, Miettinen & Nurminen Method; Difference in Percentage: Across Nights = 0.00, 95% CI 2-sided [-6.4 to 6.4]

9. Secondary Outcome: Percentage of Participants With Rebound As Defined By Decreased Subjective Total Sleep Time (sTST) During the DB Run-Out Phase
Description: Rebound insomnia was defined as insomnia that occurred following discontinuation of a sedative substance taken to relieve primary insomnia, and was assessed based on subjective total sleep time (sTST) as recorded in the participant's morning e-diary. A strict categorical analysis method (Yes/No) was used in which a participant was considered to have potentially experienced rebound (Yes) if the Morning Diary participant-reported sTST value (in minutes) on any of the 3 nights of the Run-out Phase (first 3 nights of the Discontinuation Phase) occurring after one year of treatment (Month 13) was less than the last value at baseline one year earlier (Month 1).
Time Frame: Baseline (Month 1) and first 3 days of Randomized Discontinuation Phase (otherwise known as the Run-out, Month 13)
Population: Participants in the APaT population who completed the entire DB Treatment Phase, had a baseline measurement, had taken at least one dose of DB Run-out study medication, and had a measurement on at least one of the nights of the DB Run-out Phase.
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation)
Number analyzed (Participants) | 152 | 157 | 152
percentage of participants
  Rebound on Night 1 (n=137, 142, 139) | 17.5 | 33.8 | 28.8
  Rebound on Night 2 (n=138, 146, 145) | 19.6 | 35.6 | 26.9
  Rebound on Night 3 (n=131, 146, 139) | 16.8 | 37.7 | 31.7
  Rebound on Nights 1, 2 or 3 (n=152, 157, 152) | 28.9 | 51.0 | 40.1
Statistical Analysis 1: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTST rebound effects during Night 1 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.365, Miettinen & Nurminen Method; Difference in Percentage: Night 1 = 5.03, 95% CI 2-sided [-5.8 to 15.8]
Statistical Analysis 2: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTST rebound effects during Night 2 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.109, Miettinen & Nurminen Method; Difference in Percentage: Night 2 = 8.72, 95% CI 2-sided [-2.0 to 19.2]
Statistical Analysis 3: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTST rebound effects during Night 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.287, Miettinen & Nurminen Method; Difference in Percentage: Night 3 = 6.02, 95% CI 2-sided [-5.1 to 16.9]
Statistical Analysis 4: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTST rebound effects during Nights 1, 2, or 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.057, Miettinen & Nurminen Method; Difference in Percentage:Night 1, 2 or 3 = 10.82, 95% CI 2-sided [-0.3 to 21.7]

10. Secondary Outcome: Percentage of Participants With Rebound As Defined By Increased Subjective Time to Sleep Onset (sTSO) During the DB Run-Out Phase
Description: Rebound insomnia was defined as insomnia that occurred following discontinuation of a sedative substance taken to relieve primary insomnia, and was assessed based on subjective time to sleep onset (sTSO) as recorded in the participant's morning e-diary. A strict categorical analysis method (Yes/No) was used in which a participant was considered to have potentially experienced rebound (Yes) if the Morning Diary participant-reported sTSO value (in minutes) on any of the first 3 nights of the Run-out Phase occurring after one year of treatment (Month 13) was greater than the last value at baseline one year earlier (Month 1).
Time Frame: Baseline (Month 1) and first 3 days of Randomized Discontinuation Phase (otherwise known as the Run-out, Month 13)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation)
Number analyzed (Participants) | 152 | 157 | 152
percentage of participants
  Rebound on Night 1 (n=137, 142, 139) | 16.8 | 26.8 | 22.3
  Rebound on Night 2 (n=138, 146, 145) | 18.8 | 30.1 | 24.8
  Rebound on Night 3 (n=131, 146, 139) | 19.1 | 30.1 | 25.2
  Rebound on Nights 1, 2 or 3 (n=152, 157, 152) | 31.6 | 40.8 | 36.2
Statistical Analysis 1: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTSO rebound effects during Night 1 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.386, Miettinen & Nurminen Method; Difference in Percentage: Night 1 = 4.46, 95% CI 2-sided [-5.7 to 14.5]
Statistical Analysis 2: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTSO rebound effects during Night 2 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.311, Miettinen & Nurminen Method; Difference in Percentage: Night 2 = 5.31, 95% CI 2-sided [-5.0 to 15.5]
Statistical Analysis 3: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTSO rebound effects during Night 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.351, Miettinen & Nurminen Method; Difference in Percentage: Night 3 = 4.96, 95% CI 2-sided [-5.5 to 15.3]
Statistical Analysis 4: Comparison: Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) vs Placebo (DB Treatment)/Placebo (DB Discontinuation); The method of Miettinen and Nurminen was used to calculate the p-value and compute the confidence interval for the point difference in a pairwise comparison of the percentage of participants with sTSO rebound effects during Nights 1, 2, or 3 in the Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) group vs. the Placebo (DB Treatment)/Placebo (DB Discontinuation) group; Test type: Superiority or Other; p = 0.409, Miettinen & Nurminen Method; Difference in Percentage:Night 1, 2 or 3 = 4.58, 95% CI 2-sided [-6.3 to 15.3]

11. Secondary Outcome: Least Squares (LS) Mean Change From Baseline in Mean Subjective Total Sleep Time (sTSTm) During First Month of Treatment Phase
Description: The sTSTm was defined as the average over time of daily e-diary values for a participant's report of the total amount of time spent asleep before waking for the day (measured in minutes). Weekly sTSTm values (Week 1, Week 2, etc.) were the average of the daily e-diary values for the week. A summary value of this measure for Month 1 was obtained by taking the average of weekly sTSTm values for Weeks 1 through 4; (Week 1 + Week 2 + Week 3 + Week 4) ÷ 4. LS Mean Change from Baseline in sTSTm was then calculated at Week 1, Week 2, Week 3, Week 4, and Month 1.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: Full Analysis Set (FAS)-Efficacy; all randomized participants who had ≥1 post-randomization observation for the analysis endpoint subsequent to ≥1 dose of study treatment, and baseline data for those analyses that required baseline data. The number included in the FAS may vary across endpoints due to the degree of missing data for each endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 517 | 254
minutes
  Change From BL at Week 1 (N=508, 252) | 41.1 [36.9 to 45.3] | 14.1 [8.2 to 20.1]
  Change From BL at Week 2 (N=495, 248) | 32.4 [28.1 to 36.7] | 14.7 [8.6 to 20.8]
  Change From BL at Week 3 (N=488, 241) | 39.6 [35.3 to 44.0] | 16.4 [10.3 to 22.6]
  Change From BL at Week 4 (N=473, 238) | 41.6 [37.1 to 46.1] | 18.7 [12.3 to 25.1]
  Change From BL at Month 1 Average (N=517, 254) | 38.7 [35.0 to 42.3] | 16.0 [10.8 to 21.2]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; A Longitudinal Data Analysis Model was used to test the difference in LS mean change from baseline in sTSTm for Month 1 (Average of Weeks 1, 2, 3, 4) in the Suvorexant group vs. the Placebo group; Test type: Superiority or Other; p < 0.0001, Longitudinal Data Analysis — To account for multiplicity, Hochberg's procedure was used to control the overall Type I error rate at the 5% level; Difference in LS Means: Month 1 = 22.7, 95% CI 2-sided [16.4 to 29.0]

12. Secondary Outcome: Least Squares (LS) Mean Change From Baseline in Mean Subjective Time To Sleep Onset (sTSOm) During First Month of Treatment Phase
Description: The sTSOm was defined as the average over time of daily e-diary values for a participant's report of the time he or she required to fall asleep (measured in minutes). Weekly sTSOm values (Week 1, Week 2, etc.) were the average of the daily e-diary values for the week. A summary value of this measure for Month 1 was obtained by taking the average of weekly sTSTm values for Weeks 1 through 4; (Week 1 + Week 2 + Week 3 + Week 4) ÷ 4. LS Mean Change from Baseline in sTSOm was then calculated at Week 1, Week 2, Week 3, Week 4, and Month 1.
Time Frame: Baseline, Week 1, Week 2, Week 3, and Week 4
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 517 | 254
minutes
  Change From BL at Week 1 (N=508, 252) | -17.7 [-20.9 to -14.5] | -6.8 [-11.4 to -2.3]
  Change From BL at Week 2 (N=495, 248) | -15.7 [-19.2 to -12.2] | -7.5 [-12.4 to -2.6]
  Change From BL at Week 3 (N=488, 241) | -18.7 [-22.2 to -15.2] | -10.0 [-14.9 to -5.0]
  Change From BL at Week 4 (N=473, 238) | -19.9 [-23.1 to -16.6] | -9.4 [-14.1 to -4.8]
  Change From BL at Month 1 Average (N=517, 254) | -18.0 [-20.9 to -15.1] | -8.4 [-12.5 to -4.3]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; A Longitudinal Data Analysis Model was used to test the difference in LS mean change from baseline in sTSOm for Month 1 (Average of Weeks 1, 2, 3, 4) in the Suvorexant group vs. the Placebo group; Test type: Superiority or Other; p = 0.0002, Longitudinal Data Analysis — To account for multiplicity, Hochberg's procedure was used to control the overall Type I error rate at the 5% level; Difference in LS Means: Month 1 = -9.5, 95% CI 2-sided [-14.6 to -4.5]

13. Other Pre Specified Outcome: Number of Participants Who Reported Suicidal Ideation and/or Behavior On Study Based on Responses to the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Suicidal ideation and/or behavior that occurred on study was also assessed using the C-SSRS, a rater-administered questionnaire used to prospectively assess suicidal ideation and suicidal behavior. C-SSRS assessment was based upon a clinician's interpretation of the participant's responses to the C-SSRS questions, not by a numbered scale.
  Suicidal ideation and/or behaviors identified on the C-SSRS may not have been considered an adverse event, based on the investigator's judgment.
Time Frame: From the first day of study treatment through study follow-up (up to 14 months)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Suvorexant: After a 1-week single-blind placebo run-in, participants received suvorexant (40 mg for participants aged 18 to <65 years; and 30 mg for participants aged ≥65 years) daily before bedtime for 12 months during the double-blind (DB) Treatment Phase. Following the Treatment Phase, these participants were randomized (at baseline) to suvorexant or placebo during the 2-month Randomized Discontinuation Phase.
- Placebo: After a 1-week single-blind placebo run-in, participants received dose-matched placebo to suvorexant (administered according to age) daily before bedtime for 12 months during the DB Treatment Phase. Following the Treatment Phase, these participants continued on placebo during the 2-month Randomized Discontinuation Phase.
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 521 | 258
participants | 6 | 0

ADVERSE EVENTS:
Time Frame: AEs were monitored from the time of the Prestudy Visit (~Study Day -14) up to the completion of the Follow-up call, occurring 14 days after Randomized Discontinuation Phase (~Study Day 420) or after the last dose of medication, whichever point was later.
Groups:
- Suvorexant (DB Treatment)/Suvorexant (DB Run-out)/Follow-up: Following treatment with suvorexant during both the 12-Month DB Treatment Period and the DB Run-out period, participants entered a Follow-up Phase which concluded with a follow-up phone call 14 days after the last dose of study medication (or 14 days after the Discontinuation visit, whichever time point was later) to report AEs.
- Suvorexant (DB Treatment)/Placebo (DB Run-out)/Follow-up: Following treatment with suvorexant during the 12-Month DB Treatment Period and treatment with dose-matched placebo during the DB the Run-out period, participants entered a Follow-up Phase which concluded with a follow-up phone call 14 days after the last dose of study medication (or 14 days after the Discontinuation visit, whichever time point was later) to report AEs.
- Placebo (DB Treatment)/Placebo (DB Run-out)/Follow-up: Following treatment with dose-matched placebo during both the 12-Month DB Treatment Period and the DB Run-out period, participants entered a Follow-up Phase which concluded with a follow-up phone call 14 days after the last dose of study medication (or 14 days after the Discontinuation visit, whichever time point was later) to report AEs.
Arm/Group | Suvorexant | Placebo | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) | Placebo (DB Treatment)/Placebo (DB Discontinuation) | Suvorexant (DB Treatment)/Suvorexant (DB Run-out)/Follow-up | Suvorexant (DB Treatment)/Placebo (DB Run-out)/Follow-up | Placebo (DB Treatment)/Placebo (DB Run-out)/Follow-up
Serious Adverse Events (participants affected / at risk) | 27/521 | 17/258 | 3/156 | 1/166 | 1/162 | 1/260 | 0/261 | 2/258
Other Adverse Events (participants affected / at risk) | 184/521 | 63/258 | 7/156 | 5/166 | 9/162 | 2/260 | 1/261 | 2/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=521) | Placebo (N=258) | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) (N=156) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) (N=166) | Placebo (DB Treatment)/Placebo (DB Discontinuation) (N=162) | Suvorexant (DB Treatment)/Suvorexant (DB Run-out)/Follow-up (N=260) | Suvorexant (DB Treatment)/Placebo (DB Run-out)/Follow-up (N=261) | Placebo (DB Treatment)/Placebo (DB Run-out)/Follow-up (N=258)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=521) | Placebo (N=258) | Suvorexant (DB Treatment)/Suvorexant (DB Discontinuation) (N=156) | Suvorexant (DB Treatment)/Placebo (DB Discontinuation) (N=166) | Placebo (DB Treatment)/Placebo (DB Discontinuation) (N=162) | Suvorexant (DB Treatment)/Suvorexant (DB Run-out)/Follow-up (N=260) | Suvorexant (DB Treatment)/Placebo (DB Run-out)/Follow-up (N=261) | Placebo (DB Treatment)/Placebo (DB Run-out)/Follow-up (N=258)
Fatigue (General disorders) | 34 (40) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 42 (53) | 20 (25) | 5 (5) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 28 (32) | 11 (13) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 24 (29) | 16 (19) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 43 (66) | 22 (25) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 69 (76) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.